CLINICAL TRIAL: NCT02758808
Title: Pulmonary Fibrosis Foundation Patient Registry
Acronym: PFFR
Status: Completed | Type: Observational
Sponsor: Pulmonary Fibrosis Foundation (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Kevin Flaherty, MD, MS, Chief Medical Officer, Pulmonary Fibrosis Foundation
Other Study IDs: PFF01
Record Dates: First submitted 2016-04-14; First posted 2016-05-03 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Interstitial Lung Disease (ILD); Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — whole blood, plasma, PAXgene
Oversight: Data Monitoring Committee: No

SUMMARY:
The Pulmonary Fibrosis Foundation Patient Registry will collect data on at least 2,000 patients with interstitial lung disease (ILD) at approximately 40 clinical sites in the US. The Registry is targeting enrollment of approximately 60% of the 2,000 ILD participants to have idiopathic pulmonary fibrosis (IPF). The aim of the Registry is to create a cohort of well-characterized patients with interstitial lung disease (ILD) for participation in retrospective and prospective research

DETAILED DESCRIPTION:
The Pulmonary Fibrosis Foundation Patient Registry will collect data on at least 2,000 patients with interstitial lung disease (ILD) at approximately 40 clinical sites in the US. The Registry is targeting enrollment of approximately 60% of the 2,000 ILD participants to have idiopathic pulmonary fibrosis (IPF). The aim of the Registry is to create a cohort of well-characterized patients with interstitial lung disease (ILD) for participation in retrospective and prospective research.

Patients who meet inclusion and exclusion criteria and are being treated at a Registry site can be asked to participate. Patients will be required to read and sign an Institutional review board(IRB)-approved informed consent document prior to any Registry activity taking place.

At the time of informed consent, participants will be asked to indicate if they are interested in being contacted by Registry site personnel for potential participation in future clinical trials and/or studies. Participants who opt out will not be contacted for future studies.

No clinical procedures, testing, or diagnostics will be required by virtue of Registry participation. Participants will permit Registry staff to abstract clinical data obtained as part of routine clinical care in the diagnosis and treatment of ILD. These data will be entered into a web-based, electronic data capture (EDC) by the Registry staff to at regular intervals. Some of these data will be retrospective, having been collected prior to consenting for the Registry.

Computed tomography (CT) images collected for diagnosis and / or treatment will be de-identified at the Registry site and uploaded to a secure server that is a 21 Code of Federal Regulations (CFR) Part 11, Good Clinical Practice (GCP), and HIPAA compliant online imaging repository.

Participants will be asked to complete patient reported outcome (PRO) surveys related to ILD symptoms and quality of life at the time of enrollment and during clinical follow-up visits.Participants who are not seen for clinical follow-up within 12 months will be contacted by telephone or mail by Registry site personnel to complete the PRO measures.

The University of Michigan Statistical Analysis of Biomedical and Educational Research (SABER) unit will serve as the Registry Data Coordinating Center and will manage data entered into a web based, CFR 21 Part 11 compliant electronic data capture (EDC) system by the Registry sites.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Understand and sign the informed consent document
3. ILD Diagnosis must be made / confirmed at a participating Registry center.

   1. The diagnostic evaluation must include, at a minimum, a medical history, physical examination, pulmonary function testing and a computerized tomography (CT) scan of the chest.
   2. If patients exhibit another pulmonary disease (such as emphysema or asthma), the primary disease must be ILD.
4. Anticipated additional follow up at the Registry center within one year.

Exclusion Criteria:

1. Diagnosed with:

1. Sarcoid
2. Lymphangioleiomyomatosis (LAM)
3. Pulmonary alveolar proteinosis (PAP)
4. Cystic fibrosis (CF)
5. Amyloidosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 2,000 patients with interstitial lung disease (ILD) at approximately 40 clinical sites in the US. The Pulmonary Fibrosis Foundation Patient Registry will collect data on at least 2,000 patients at approximately 40 clinical sites in the US. The Registry is targeting enrollment of approximately 60% of the 2,000 ILD participants to have idiopathic pulmonary fibrosos (IPF).
Sampling Method: Non-Probability Sample
Enrollment: 2004 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Change in % predicted FVC | Up to 55 months
  Analysis of registry data will lead to aggregated reports summarizing the pulmonary function
Change in % predicted DLCO | Up to 55 months
  Analysis of registry data will lead to aggregated reports summarizing the pulmonary function

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Flaherty, MD, Study Chair — University of Michigan
Locations (42):
- United States (42):
  - University fo Alabama at Birmingham, Birmingham, Alabama
  - Dignity Health St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - The University of Arizona, Tucson, Arizona
  - UCLA, David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - National Jewish Health, Denver, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Piedmont Healthcare, Austell, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University - School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Regents of the University of Minnesota Twin Cities, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Health System, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - UTHSC - San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Interstitial Lung Disease Clinic, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adegunsoye A, Bachman WM, Flaherty KR, Li Z, Gupta S. Use of Race-Specific Equations in Pulmonary Function Tests Impedes Potential Eligibility for Care and Treatment of Pulmonary Fibrosis. Ann Am Thorac Soc. 2024 Aug;21(8):1156-1165. doi: 10.1513/AnnalsATS.202309-797OC. PMID 38386005
- [Derived] Lee JS, Martin-Schwarze A, Freiheit E, Trzaskoma B, Burg C. Real-World Clinical Outcomes Based on Body Mass Index and Annualized Weight Change in Patients with Idiopathic Pulmonary Fibrosis. Adv Ther. 2023 Feb;40(2):691-704. doi: 10.1007/s12325-022-02382-0. Epub 2022 Dec 8. PMID 36481866